CLINICAL TRIAL: NCT05567042
Title: A Clinical Study of Epilepsy Localization and Prognosis Based on Positron Emission Tomography and Resting-state Functional Magnetic Resonance Imaging
Brief Title: A Clinical Study of Epilepsy Localization and Prognosis Based on PET and Resting-state fMRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Li Shuangshuang (Other)
Responsible Party: Sponsor-Investigator, Li Shuangshuang, Principal Investigator, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: 20222137
Record Dates: First submitted 2022-09-26; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Epileptic Seizure
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- drug-resistant epilepsy: No intervention
  Interventions: Other: No intervention
- Medication is effective: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
1. By following up the prognosis of surgical patients, the application value of Cortex ID quantitative analysis in the localization of epilepsy foci was studied.
2. By studying the correlation between autonomic nerve function and epilepsy neural network in epilepsy patients, and analyzing the differences between different epilepsy patients, it can provide more information for judging the prognosis of epilepsy patients.

DETAILED DESCRIPTION:
This study included diagnostic trials and case-control studies, which were observational studies with no intervention. First, the demographic and clinical information of epilepsy patients in the Neurology Department of Xijing Hospital were collected, including gender, age, age of onset, course of epilepsy, seizure performance before treatment, seizure frequency before treatment, type and dose of antiepileptic drugs, past history, Family history, etc., as well as imaging, EEG, quality of life, and neuropsychological assessment, etc. were collected; secondly, functional magnetic resonance imaging (fMRI) and 24-hour Holter monitoring were performed on patients who met the inclusion criteria. Positron Emission Computed Tomography (PET) images of patients who have undergone or plan to undergo surgery are analyzed; finally, appropriate statistical methods are used for analysis.

ELIGIBILITY:
Inclusion Criteria:

Meet the diagnostic criteria for epilepsy,

* No contraindications for fMRI examination.
* The patient had no other heart and lung diseases except epilepsy.
* Patients and their families were aware of this study and signed informed consent.

Exclusion Criteria:

* Patients with severe infection, cerebrovascular disease, malignant tumor and other systemic diseases that can affect the nervous system, and those with serious dysfunction of the heart, liver, kidney and other organs.
* Non-epileptic seizures such as syncope and hysteria.
* Pregnant or lactating women. Incomplete clinical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational study of epilepsy patients treated at the Epilepsy Center of Xijing Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | 2022-2024
Seizure duration | 2022-2024

IPD SHARING:
Plan to Share IPD: Undecided
Make decisions based on research progress

REFERENCES:
- [Background] Kassinopoulos M, Harper RM, Guye M, Lemieux L, Diehl B. Altered Relationship Between Heart Rate Variability and fMRI-Based Functional Connectivity in People With Epilepsy. Front Neurol. 2021 Jun 10;12:671890. doi: 10.3389/fneur.2021.671890. eCollection 2021. PMID 34177777